CLINICAL TRIAL: NCT00246415
Title: Medications Development for Alcohol Abuse: NMDA Agents -- A Placebo-Controlled Trial of Memantine for Alcohol Dependence
Brief Title: A Placebo-Controlled Trial of Memantine for Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAA-EVA12599; NIH RO1 AA12599
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Alcohol Dependence (Primary Condition); Alcohol Abuse
Keywords: Alcohol Dependence; Alcohol Abuse; Memantine; Alcohol Treatment
MeSH Terms: conditions — Alcoholism | interventions — Memantine

INTERVENTIONS:
Drug: Memantine

SUMMARY:
The purpose of this study is to obtain a preliminary indication of the safety and effectiveness of oral memantine (40 mg/day) in alcohol dependent patients. This study is a 16-week study comparison of memantine and placebo in patients with alcohol dependence.

DETAILED DESCRIPTION:
This study is a 16-week study, double-blind, parallel groups, two arm comparison of memantine and placebo in patients with alcohol dependence.

Procedures. This outpatient clinical trial comprises a 2-week placebo lead-in phase followed by a 12-week treatment phase and a 2-week lead-out phase. Patients will be seen 2x/week. There will also be a 3-month follow-up visit to reassess the status of abstinence or relapse to drinking. The design of the study is as follows:

Single-blind Placebo Lead-in Phase (Week -2 and Week -1). Patients who give informed consent and provisionally meet the inclusion-exclusion criteria will enter a 2-week Single-blind Placebo Lead-in Phase. After this placebo lead-in phase, patients will be randomized to receive memantine or placebo and they will be stratified by sex, age, race and level of alcohol dependence.

12 Week Treatment Phase (Weeks 1-12). At these visits, medication will be provided, standardized assessment instruments will be completed, and biochemical measures will be taken to monitor alcohol consumption as well as compliance with study medication. In one of these two weekly visits patients will receive individual, manual-guided relapse prevention therapy with a clinician and meet with a study psychiatrist. Patients wishing to take naltrexone (ReVia), disulfiram (Antabuse), or participate in more intensive inpatient treatment during the trial will be discontinued from the study.

Single-blind Lead-out Phase (Weeks 13-14). During this 2-week lead-out phase, patients on active medication will be tapered off the medication to placebo, but all other measures and assessments (including weekly psychotherapy sessions) will remain the same. All patients, regardless of whether they complete the study or are administratively removed, will be followed up and rated at Week 14. There will also be a 3-month follow-up visit to reassess the status of abstinence or relapse to drinking.

Clinic Visits. During these visits, the research nurse and a research assistant measure breath alcohol content (BAC), urine and blood samples as scheduled for monitoring alcohol, illicit drug use, and medication compliance. Medication compliance will initially be assessed by measuring riboflavin fluorescence in urine samples. The staff will supervise the completion of self-report questionnaires. The nurse will check vital signs at each visit, weight once per week and will question patients about compliance, any missed doses, and possible side effect or other adverse events, and will complete the compliance and adverse events forms. Medication compliance will be monitored via riboflavin (Del Boca et al 1996), self-report data, collateral informant data, and medication blood levels. Likewise, drinking behavior will be monitored with BAC, self-report and collateral informant data. This data will be available to the treatment team and will be used to reinforce importance of compliance. The patient will meet weekly with the psychiatrist who will assess current alcohol use and mood status, evaluate side effects and adjust dosage as needed (using the prearranged blinded dose adjustment schedule), review events occurring since the last study visit relating to the patient's functioning, and perform the CGI-Observer rating. During one of the two weekly visits, the patient will also meet with the therapist for individual relapse prevention therapy. At any point during the trial, if the treating psychiatrist determines that the primary alcohol dependence, secondary dependence on other drugs of abuse, or new drug dependence has escalated such that a more intensive intervention is required, he/she will make decisions about removal from the trial and referral to other forms of treatment.

Medication will be given on a fixed-flexible schedule, titrated to the maximum recommended dose to minimize side effects. Patients will receive enough medication to last until the next visit. For patients assigned to memantine, they will be gradually titrated from 10 mg/day to the maximal dose of 20 mg b.i.d. (40 mg/day) over the first two weeks of the treatment phase. All patients will receive matching pills in the same quantity each day. In case of several missed visits, side effects or adverse events, a study nurse and a study psychiatrist will meet with the patient and a dose decrease will be arranged using the prearranged blinded dose adjustment schedule. Patients who cannot tolerate 50% of the maximal dose (i.e., 20 mg/day memantine) will be discontinued from study medication; however, based on our experience, this is highly unlikely.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18-65 yrs.
2. Meets DSM-IV criteria for current alcohol dependence. Volunteers may meet criteria for other substance abuse, or dependence on other drugs (nicotine, marijuana or cocaine) as long as the dependence on marijuana or cocaine is secondary to alcohol dependence
3. Medically healthy on the basis of physical examination and medical history, vital signs, ECG and laboratory tests, with a negative blood pregnancy test for females.
4. Expresses desire to stop drinking alcohol.
5. Does not require any psychotropic medication.
6. Able to provide informed consent and comply with study procedures.
7. Signed informed consent.

Exclusion Criteria:

1. Dependence on opiates
2. Meets DSM-IV criteria for schizophrenia or bipolar Disorder. Has a psychotic illness or is at risk for suicidal behavior.
3. History of delerium tremens (hallucinations, psychosis, agitation) secondary to alcohol withdrawal, a personal or family history of seizure disorder, a personal history of moderate/severe head trauma.
4. Currently taking psychotropic medication.
5. In need of inpatient alcohol detoxification.
6. Any renal disease or insufficiency.
7. Clinically significant and symptomatic medical disorder requiring active intervention
8. Female patients who are lactating or who have childbearing potential and who refuse to use birth control (hormone or barrier) or are pregnant.
9. Patients for whom treatment of alcoholism is being mandated by legal action.
10. Patients with active malignancy (other than non- melanoma skin cancer of carcinoma in situ of uterine cervix) within 5 years of beginning study.
11. Known or suspected hypersensitivity to memantine.
12. Intolerable adverse event during Single Blind Placebo Lead-in Phase.
13. Patients taking naltrexone or antabuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2002-11; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption- Standard Drink Units (Time line Followback)
Abstinence from alcohol (Time line Followback)

SECONDARY OUTCOMES:
Clinical Global Impression-Alcohol

CONTACTS AND LOCATIONS:
Overall Officials: Suzette M. Evans, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Risnes LF, Eggesbo LM, Zuhlke S, Dahal-Koirala S, Neumann RS, Lundin KEA, Christophersen A, Sollid LM. Circulating CD103+ gammadelta and CD8+ T cells are clonally shared with tissue-resident intraepithelial lymphocytes in celiac disease. Mucosal Immunol. 2021 Jul;14(4):842-851. doi: 10.1038/s41385-021-00385-8. Epub 2021 Mar 2. PMID 33654213